CLINICAL TRIAL: NCT06553716
Title: Ultrasound-Guided Hydrodilatation With Triamcinolone Acetonide for Adhesive Capsulitis:The Effect of the Rotator Cuff Interval With Posterior Glenohumeral Recess Approaches on the Improvement of Joint Motion and Pain
Brief Title: Ultrasound-Guided Hydrodilatation With Triamcinolone Acetonide for Adhesive Capsulitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Peng Ma-2024-0201
Record Dates: First submitted 2024-08-11; First posted 2024-08-14 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Postoperation Pain
Keywords: Adhesive capsulitis; hydrodilatation; corticosteroid; rotator cuff interval; Posterior Glenohumeral Recess
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rotator cuff space approach (GroupA) (Active Comparator): In the Rotator cuff interval recess group,we injected 20 mL lidocaine with 2 mg/mL triamcinolone acetonide (Shincort) into into the Rotator cuff interval/anterior capsule.
  Interventions: Procedure: Ultrasound-Guided Hydrodilatation by the Rotator cuff interval recess
- Rotator cuff space approach combined with posterior glenohumeral recess approach (GroupB) (Experimental): In the Rotator cuff interval and posterior glenohumeral recess group,we injected 10 mL lidocaine with 2 mg/mL triamcinolone acetonide (Shincort) into the Rotator cuff interval/anterior capsule and 10 mL mL lidocaine with 2 mg/mL triamcinolone acetonide (Shincort) into the posterior glenohumeral.
  Interventions: Procedure: Ultrasound-Guided Hydrodilatation by the Rotator cuff interval and posterior glenohumeral recess

INTERVENTIONS:
Procedure: Ultrasound-Guided Hydrodilatation by the Rotator cuff interval recess — The injection contained 5ml of triamcinolone acetonide (40 mg)mixed with 5ml of 2% lidocaine hydrochloride and 15ml of normal saline in both groups,In the Rotator cuff interval recess group,we injected 20 mL lidocaine with 2 mg/mL triamcinolone acetonide (Shincort) into into the Rotator cuff interval/anterior capsule.
  Arms: Rotator cuff space approach (GroupA)
Procedure: Ultrasound-Guided Hydrodilatation by the Rotator cuff interval and posterior glenohumeral recess — The injection contained 5ml of triamcinolone acetonide (40 mg)mixed with 5ml of 2% lidocaine hydrochloride and 15ml of normal saline in both groups,In the Rotator cuff interval and posterior glenohumeral recess group,we injected 10 mL lidocaine with 2 mg/mL triamcinolone acetonide (Shincort) into the Rotator cuff interval/anterior capsule and 10 mL mL lidocaine with 2 mg/mL triamcinolone acetonide (Shincort) into the posterior glenohumeral.
  Arms: Rotator cuff space approach combined with posterior glenohumeral recess approach (GroupB)

SUMMARY:
The purpose of this study was to compare the efficacy of ultrasus-guided hydrodilation of Rotator Cuff Interval combined with Posterior Glenohumeral recess approach and hydrodilation of the Rotator cuff Interval alone in Adhesive Capsulitis.

DETAILED DESCRIPTION:
For patients with perihumeral arthritis, shoulder capsule hydrodilation is usually performed using ultrasound-guided water dilation through the posterior glenohumeral recess. Recently, a new transrotator cuff space approach has been described, and this study was designed to compare the efficacy of triamcinolone olonide transrotator cuff space combined with posterior glenohumeral recess and rotator cuff space dilation in the treatment of adhesive joint capsitis.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, clinical diagnosis of periarthritis of shoulder;
2. symptom duration > 1 month, shoulder ROM limitation in at least two directions, defined as abduction < 80°, flexion < 130°, and rotation < 30°;
3. Before enrollment, the patients received plain radiographs, ultrasound images, and magnetic resonance imaging to rule out the cause of secondary shoulder capsitis.

Exclusion Criteria:

1. Secondary frozen shoulder, such as rotator cuff tear, calcifying tendinitis, osteoarthritis, infection, tuberculosis infection, rheumatic disease, shoulder impingement syndrome;
2. Previous history of shoulder joint surgery;
3. Involved cervical nervous system symptoms or abnormal nervous system;
4. corticosteroid injection in the affected shoulder within 3 months;
5. Mental illness;
6. Patients with contraindications to cortisol-hormone use.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Shoulder Pain and Disability Index | At baseline, one week, three weeks, six weeks, 12 weeks after treatment.
  The SPADI was used to assess the severity ofpain and disability. A previous study has shown that the Chinese version of the SPADI has high internal consistency and test-retest reliability (Yao et al., 2017). It consists of 13 items that are divided into 2 subscales: pain scale (5 items) and disability scale (8 items) (Roach et al., 1991). Each item is rated from 0 (no pain/no difficulty) to 10 (worst pain experienced/ very difficult). The score is then transformed to a 100-point scale, with the highest score indicating the most severe pain and disability. In the literature, the minimal and clinically relevant difference for SPADI has been reported to be 10 points

SECONDARY OUTCOMES:
visual analogue scale | At baseline, one week, three weeks, six weeks, 12 weeks after treatment.
  Regarding VAS, patients were asked to indicate the intensity of their average level ofpain in the affected shoulder within the past 1 week using an 11-point scale, ranging from 0 (no pain) to 10 (worst pain imaginable).
Active shoulder range of motion | Baseline data, six weeks,12 weeks after treatment
  In terms of ROM, the degrees of shoulder flexion, abduction, external and internal rotation were measured by a goniometer in the supine position in a random sequence
adverse reaction | one week after treatment
  Pain after hydrodilation , reduced sensation and motor control of the affected arm, skin flushing, nausea, dizziness, and fainting

CONTACTS AND LOCATIONS:
Locations (1):
- General hospital of Ningxia medical university, Yinchuan, Ningxia, China

IPD SHARING:
Plan to Share IPD: No